CLINICAL TRIAL: NCT02429583
Title: Effects of Persistent Innate Immune Activation on Vaccine Efficacy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll sufficient subjects
Sponsor: Rockefeller University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Charles Rice, Head of Laboratory of Virology and Infectious Disease, Rockefeller University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CRI-0844; U19AI111825 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — Recombivax HB; Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recombivax in HCV infected individuals (Active Comparator): Recombivax vaccine administered IM to HCV-infected individuals
  Interventions: Drug: Recombivax
- Recombivax in healthy volunteers (Active Comparator): Recombivax vaccine administered IM to healthy individuals
  Interventions: Drug: Recombivax

INTERVENTIONS:
Drug: Recombivax — Injection of Recombivax HBV vaccine administered IM, at 0, 1, and 6 months after enrollment
  Other Names: Hepatitis B vaccine

SUMMARY:
This study will investigate the effects of chronic HCV infection and corresponding innate immune activation on the immune response to HBV vaccination. We will recruit chronic HCV patients and healthy control patients for HBV vaccination. We will use RNA Sequencing (RNA-Seq), a relatively new technology for simultaneously measuring the expression of all genes, to determine patients' innate immune status, and learn how this innate immune signature is related to HBV vaccine response. We will then explore the mechanisms by which chronic HCV infection affects different immune cells and functions that are known to be important for an effective HBV vaccine response. These studies will enhance our understanding of the immune effects of chronic viral infection, establish factors that determine effective vaccine responses, and help guide vaccination strategies for HCV patients and other individuals with chronic inflammatory disease.

DETAILED DESCRIPTION:
Vaccines have been responsible for preventing millions of deaths and extending the average human lifespan. Effective vaccines stimulate the cells of the immune system to activate genes and associated functions that bring about protective immunity. If we can better understand the factors that influence vaccine success versus failure, we may be able to improve current vaccines and/or develop new vaccines against prevalent infectious diseases.

Certain groups of people do not respond well to particular vaccines. For example, vaccines can be less effective in immunocompromised patients, elderly individuals, and people with chronic inflammatory diseases. Often it is these groups of people that have the greatest need for protection against infectious disease.

People chronically infected with hepatitis C virus (HCV) are at increased risk of serious liver disease. As a result, they should receive the hepatitis B virus (HBV) vaccine, which can protect them from infection by HBV, another virus that targets the liver. However, people chronically infected with HCV do not respond to the HBV vaccine as effectively as healthy people without HCV. Chronic HCV infection is not thought to cause general problems with the immune system, and the reasons for this poor vaccine response are poorly understood. Previous work has shown that chronic HCV infection leads to production of chemical ("innate immune") signals that can affect function of the immune system, but it is currently unknown how this might impact vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Willing to receive three doses of an FDA-approved Hepatitis B vaccine
* Volunteer chronically infected with HCV (as demonstrated by serology and/or viral load laboratory studies)
* Healthy volunteer without significant medical problems

Exclusion Criteria:

* Received any vaccine within a month prior to study vaccine
* Positive serum antibody against Hep B surface antigen and/or core Hep B core antigen
* HIV positive
* For HCV-negative, healthy volunteers: History of HCV infection or positive HCV antibody test
* Participation in another clinical study of an investigational product currently or within the past 90 days, or expected participation during this study
* In the opinion of the investigator, the volunteer is unlikely to comply with the study protocol
* Any clinically significant abnormality or medical history or physical examination including history of immunodeficiency or autoimmune disease (in addition to HCV infection, for HCV group)
* Currently taking systemic steroids or other immunomodulatory medications including anticancer medications and antiviral medications
* Any clinically significant acute or chronic medical condition requiring care by a primary care provider (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that, in the opinion of the investigator, would preclude participation
* Unable to continue participation for 156 weeks
* History of previous Hepatitis B vaccination(s)
* Male or female < 18 and > 62 years of age
* Is pregnant or lactating
* History of Hepatitis B infection
* Clinical, laboratory, or biopsy evidence of cirrhosis

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rice, PhD, Principal Investigator — The Rockefeller University Center for Clinical and Translational
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Recombivax in HCV Infected Individuals | Recombivax in Healthy Volunteers
Started | 1 | 23
Completed | 1 | 3
Not Completed | 0 | 20

BASELINE CHARACTERISTICS:
Population: Only 4 participants completed the study. One HCV infected individual enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombivax in HCV Infected Individuals | Recombivax in Healthy Volunteers | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 60 [60 to 60] | 44 [42 to 49] | 48 [42 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: HBV Vaccine Response Versus Non-response Status
Description: Titers of anti-hepatitis B surface antigen antibody measured at 8 months
  Luminex assay for multiplex cytokine/chemokine panel measured at 8 months RNA-Seq with analysis focus on curated ISG list measured at 8 months
Time Frame: 8 months
Population: The data was not collected and the analysis was not completed for this study due to insufficient enrollment.
Arm/Group | Recombivax in HCV Infected Individuals | Recombivax in Healthy Volunteers
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Frequency and Functional Status of Anti-HBsAg Antibody-producing B Cells Post-vaccination Doses Over Time
Description: ELISPOT assays will measured at 8 months
Time Frame: 8 months
Population: The data was not collected and the analysis was not completed for this study due to insufficient enrollment.
Arm/Group | Recombivax in HCV Infected Individuals | Recombivax in Healthy Volunteers
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Frequency and Functional Status of HBsAg-specific CD4+ "Helper" T Cells
Description: Flow cytometry assays measured at 8 months
Time Frame: 8 months
Population: The data was not collected and the analysis was not completed for this study due to insufficient enrollment.
Arm/Group | Recombivax in HCV Infected Individuals | Recombivax in Healthy Volunteers
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Functional Response of Monocytes Stimulated ex Vivo With Vaccine Antigen and/or Adjuvant
Description: Isolated from patient PBMCs measured at 8 months
Time Frame: 8 months
Population: The data was not collected and the analysis was not completed for this study due to insufficient enrollment.
Arm/Group | Recombivax in HCV Infected Individuals | Recombivax in Healthy Volunteers
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Gene Expression Profile of Conventional Dendritic Cells Measured by RNA-Seq
Description: Isolated from patient PBMCs measured at 8 months
Time Frame: 8 months
Population: The data was not collected and the analysis was not completed for this study due to insufficient enrollment.
Arm/Group | Recombivax in HCV Infected Individuals | Recombivax in Healthy Volunteers
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 weeks
Description: Adverse event information was collected from both arms of the study (3 healthy volunteers and 1 HCV infected individual)
Arm/Group | Recombivax in HCV Infected Individuals | Recombivax in Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombivax in HCV Infected Individuals (N=1) | Recombivax in Healthy Volunteers (N=3)
Cold Like Symptoms (General disorders) | 0 | 1 (1) — Volunteer complained of "cold-like" symptoms (headache, sneezing, scratchy throat) without cough or fever.
Patient Stubbed Toe (General disorders) | 0 | 1 (1) — Volunteer reported that he stubbed the great toe of his left foot on 08/19/2015 resulting in moderate pain and discomfort
Pain at Injection Site (Surgical and medical procedures) | 0 | 1 (1) — Volunteer experienced mild tenderness at the right upper arm vaccination site twenty minutes after receiving his first Hepatitis B vaccination which resolved by next day

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT02429583/Prot_SAP_000.pdf